CLINICAL TRIAL: NCT04605536
Title: Effect of Animation Video on the Success Rate of Children Swallowing Capsule Endoscopy: a Randomized Controlled Trial
Brief Title: Effect of Animation Video on the Success Rate of Children Swallowing Capsule Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Director, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE_swallowing
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Capsule Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Give explanations about conventional capsule endoscopy and watch animation videos
  Interventions: Other: animation videos; Other: explanation about endoscopy endoscopy
- Control (Other): Give explanations about conventional capsule endoscopy
  Interventions: Other: explanation about endoscopy endoscopy

INTERVENTIONS:
Other: animation videos — watch animation videos about capsule endoscopy
  Arms: Intervention
Other: explanation about endoscopy endoscopy — Give general explanations about endoscopy endoscopy

SUMMARY:
There are a variety of strategies that can be used for education to improve patients' awareness of the electronic capsule endoscopy process at present. The animated images in the animation videos are interesting as the explanations are simple and easy to understand. It is one of the best choices for children's education. A number of studies have shown that animated videos can increase the awareness rate of children's related knowledge, reduce anxiety, improve children's compliance with examinations and operations, and achieve good clinical results. Effective information transmission to children and their family members can increase the children's cognition and may affect the children's compliance with swallowing capsules and the success rate of autonomous swallowing, thereby reducing the time for swallowing capsule endoscopes and increasing capsule endoscopes Complete small bowel examination completion rate. This study aimed to evaluate the impact of animated video education on the success rate of children swallowing capsule endoscopy and analyze the related factors that affect the time for children to swallow capsules autonomously.

ELIGIBILITY:
Inclusion Criteria:

* Have indications for capsule endoscopy;
* Agree to undergo capsule endoscopy;
* Have normal intelligence and can communicate with the operator normally.

Exclusion Criteria:

* Contraindications for capsule endoscopy;
* Previous experience of capsule endoscopy;
* Allergic to polymer materials;
* Persons with mental retardation;
* Those who cannot communicate normally due to diseases or emotions;
* A HAMA scale of 21 or above, which indicates severe anxiety, before the examination

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
success rate of swallowing capsule endoscopy | 48 hours
  The success rate of children swallowing capsule endoscopy spontaneously

SECONDARY OUTCOMES:
HAMA anxiety score | 24 hours
  Hamilton Anxiety Scale before capsule endoscopy examination, the lowest score means the least anxiety
Swallowing time | 24 hours
  Time to swallow the capsule endoscopy
Heart rate | 48 hours
  Heart rate of children before and during the capsule endoscopy
Adverse effects | 24 hours
  Adverse effects after swallowing the capsule endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arguelles-Arias F, Donat E, Fernandez-Urien I, Alberca F, Arguelles-Martin F, Martinez MJ, Molina M, Varea V, Herrerias-Gutierrez JM, Ribes-Koninckx C. Guideline for wireless capsule endoscopy in children and adolescents: A consensus document by the SEGHNP (Spanish Society for Pediatric Gastroenterology, Hepatology, and Nutrition) and the SEPD (Spanish Society for Digestive Diseases). Rev Esp Enferm Dig. 2015 Dec;107(12):714-31. doi: 10.17235/reed.2015.3921/2015. PMID 26671584